CLINICAL TRIAL: NCT01165164
Title: An Evaluation of the Nighttime Retention of Effect of an Investigational Lubricant Eye Drop (FID 115958D)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-10-014
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye
Keywords: Dry eye; artificial tears
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Lubricant Eye Drops

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FID 115958D (Experimental): Lubricant eye drop
  Interventions: Other: FID 115958D (lubricant eye drop)

INTERVENTIONS:
Other: FID 115958D (lubricant eye drop) — 1 drop in each eye at bedtime

SUMMARY:
The purpose of this study is to describe the night-time use of an investigational lubricant eye drop.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of dry eye
2. Current use of an eye ointment or tube gel

Exclusion Criteria:

1. No nighttime contact lenses wear throughout the study period
2. Must not have had punctal plugs inserted within 30 days preceding enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Nighttime Use Assessment | Day 7
  Nighttime Use Assessment: "I would use this product at bedtime for my dry eye symptoms" Likert scale (i.e. strongly disagree, disagree, neither disagree nor agree, agree, strongly agree)